CLINICAL TRIAL: NCT06133244
Title: Hand Function Impairment in Systemic Sclerosis: Outcomes, Mechanisms and Experience (HANDSOME) Study
Brief Title: Hand Function Impairment in Systemic Sclerosis: Outcomes, Mechanisms and Experience (HANDSOME)
Status: Recruiting | Type: Observational
Sponsor: UMC Utrecht (Other)
Collaborators: University Medical Center Groningen (Other); Radboud University Medical Center (Other); Leiden University Medical Center (Other); Royal Free Hospital NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Julia Spierings, MD PhD, Dr., UMC Utrecht
Other Study IDs: NL85445.041.23
Record Dates: First submitted 2023-11-10; First posted 2023-11-15 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Systemic Sclerosis
MeSH Terms: conditions — Scleroderma, Systemic | interventions — Diagnostic Imaging; Blood Specimen Collection; Physical Examination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- VEDOSS: defined as RP, presence of SSc specific autoantibodies (ACA, ATA, ARA), puffy fingers and abnormal nailfold capillaroscopy (giant capillaries or capillary loss with or without haemorrhages), but not fulfilling the EULAR-ACR 2013 classification criteria for SSc
  Interventions: Diagnostic Test: Imaging, blood samples, fuctional tests and physical examination
- SSc with disease duration of < 4 years without hand contractures
  Interventions: Diagnostic Test: Imaging, blood samples, fuctional tests and physical examination
- SSc with hand contractures
  Interventions: Diagnostic Test: Imaging, blood samples, fuctional tests and physical examination

INTERVENTIONS:
Diagnostic Test: Imaging, blood samples, fuctional tests and physical examination — Imaging, blood samples, fuctional tests and physical examination

SUMMARY:
Almost 90% of systemic sclerosis (SSc) patients experience hand function limitation, which leads to impaired daily functioning and work participation. An important cause of impaired hand function are contractures of the hand, which are reported in up to a half of patients. With this longitudinal cohort study in patients with SSc and VEDOSS (very early diagnosis of systemic sclerosis) the investigators aim to gain more insight into processes involved in hand function impairment.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years

Exclusion Criteria:

* Patients with diabetic cheiroarthropathy and Dupuytren's disease, based on expert opinion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients (18 years and older) with:
  1. SSc with hand contractures
  2. SSc patients without contractures and disease duration of < 4 years
  3. VEDOSS patients
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-04-19 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Determination of risk factors for hand function impairment in systemic sclerosis (SSc) patients with early disease, very early disease and established hand impairment (contractures) at 2 years follow-up | 2 years

SECONDARY OUTCOMES:
Identify underlying mechanisms | 2 years
- Validation of the Dutch PASTUL questionnaire | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- UMC Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Greveling M, Ong VH, Denton C, Foppen W, Herman A, Jeffries-Owen N, Kortekaas M, Masselink I, Mulder DJ, Schriemer R, Vonk MC, de Vries-Bouwstra JK, Welsing P, Mastbergen S, Spierings J. Hand function impairment in Systemic sclerosis: Outcomes, Mechanisms and Experience (HANDSOME) - a longitudinal observational multicentre study protocol. BMJ Open. 2025 Mar 13;15(3):e095283. doi: 10.1136/bmjopen-2024-095283. PMID 40082008